CLINICAL TRIAL: NCT02582515
Title: Augmentation of Brief Habit Reversal Training With D-cycloserine or Placebo
Acronym: DCS+HRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Joseph McGuire, Postdoctoral Fellow and Clinical Instructor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCLA_DCS+HRT
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Tourette Disorder; Chronic Tic Disorder
Keywords: d-cycloserine; comprehensive behavioral intervention for tics; habit reversal training
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-cycloserine + Habit Reversal Training (Experimental): Participants randomly assigned to the D-cycloserine (DCS) condition will receive a single dose of DCS immediately prior to a single session of habit reversal training.
  Interventions: Drug: D-cycloserine
- Placebo + Habit Reversal Training (Placebo Comparator): Participants randomly assigned to the placebo condition will receive a single dose of placebo immediately prior to a single session of habit reversal training.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine
  Other Names: Habit Reversal Training
  Arms: D-cycloserine + Habit Reversal Training
Drug: Placebo
  Other Names: Habit Reversal Training
  Arms: Placebo + Habit Reversal Training

SUMMARY:
Expert reviews and practice parameter papers recommend behavior therapy as a first-line intervention for youth with chronic tic disorders (CTDs) with mild-to-moderate tic severity. Although behavior therapies like the Comprehensive Behavioral Intervention for Tics (CBIT) are efficacious in reducing tic symptom severity, only 50% of individuals exhibit a positive treatment response. Thus, there is a clear need to identify strategies to improve treatment response and/or accelerate therapeutic gains .

The primary ingredient of CBIT is habit reversal training (HRT), which utilizes both extinction and associative learning. Psychosocial treatments relying on these learning mechanisms have demonstrated an enhanced and/or expedited therapeutic benefit when augmented with d-cycloserine (DCS). This feasibility study will examine the incremental efficacy of HRT+DCS over HRT+placebo for tics targeted with HRT. Eligibility criteria will parallel the child CBIT trial for generalizability and comparability, with the addition of DCS contraindications as exclusionary criteria. Parents and youth will complete a battery of clinical assessments to ascertain tic symptoms severity and co-occurring psychiatric conditions. Afterwards, participants will be randomly assigned to receive either HRT+DCS or HRT+placebo. Instead of a full course of HRT (8 sessions over 10 weeks), a more efficient Quick-Win/Fast-Fail trial design will be used that includes a truncated HRT protocol to provide results in a more timely fashion. As a result of this trial design, the primary outcome of this study will focus on the reduction of bothersome tic severity for those targeted in treatment rather than global severity reductions.

DETAILED DESCRIPTION:
Expert reviews and practice parameter papers recommend behavior therapy as a first-line intervention for youth with chronic tic disorders (CTDs) with mild-to-moderate tic severity. Although behavior therapies like the Comprehensive Behavioral Intervention for Tics (CBIT) are efficacious in reducing tic symptom severity, only 50% of individuals exhibit a positive treatment response. Thus, there is a clear need to identify strategies to improve treatment response and/or accelerate therapeutic gains. The primary ingredient of CBIT is habit reversal training (HRT), which utilizes both extinction and associative learning. Psychosocial treatments relying on these learning mechanisms have demonstrated an enhanced and/or expedited therapeutic benefit when augmented with d-cycloserine (DCS). This feasibility study will examine the incremental efficacy of HRT+DCS over HRT+placebo for tics targeted with HRT. Eligibility criteria will parallel the child CBIT trial for generalizability and comparability, with the addition of DCS contraindications as exclusionary criteria. Parents and youth will complete a battery of clinical assessments to ascertain tic symptoms severity and co-occurring psychiatric conditions. Afterwards, participants will be randomly assigned to receive either HRT+DCS or HRT+placebo. Instead of a full course of HRT (8 sessions over 10 weeks), a more efficient Quick-Win/Fast-Fail trial design will be used that includes a truncated HRT protocol to provide results in a more timely fashion. As a result of this trial design, the primary outcome of this study will focus on the reduction of bothersome tic severity for those targeted in treatment rather than global severity reductions.

ELIGIBILITY:
Inclusion Criteria:

1. ages 8 years to 17 years (inclusive);
2. meet diagnostic criteria for either Tourette Disorder or a Persistent Tic Disorder;
3. moderate tic severity or greater as evidenced by a Yale Global Tic Severity Scale (Leckman, Riddle, Hardin, & Ort, 1989) total score greater than 13 (>9 for children with motor or vocal tics only);
4. be fluent in English;
5. be medication free or on a stable dose of a non-antipsychotic medication for 6 weeks with no planned changes.

Exclusion Criteria:

1. pregnant or breast feeding;
2. an unstable medical condition (e.g., a seizure disorder, kidney or liver disease);
3. current diagnosis of substance abuse/dependence;
4. lifetime diagnosis of schizophrenia, autism spectrum disorder, bipolar disorder, or psychosis;
5. evidence of a seizure disorder, kidney or liver disease, pregnant and/or breast feeding;
6. four or more previous sessions of HRT; or
7. currently taking an antipsychotic medication.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F McGuire, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- D-cycloserine + Habit Reversal Training: Participants randomly assigned to the D-cycloserine (DCS) condition will receive a single dose of DCS immediately prior to a single session of habit reversal training. Participants will be evaluated 1 week later for improvement in tics targeted in the treatment session.
  D-cycloserine
- Placebo + Habit Reversal Training: Participants randomly assigned to the placebo condition will receive a single dose of placebo immediately prior to a single session of habit reversal training. Participants will be evaluated 1 week later for improvement in tics targeted in the treatment session.
  Placebo
Period: Overall Study
Arm/Group | D-cycloserine + Habit Reversal Training | Placebo + Habit Reversal Training
Started | 9 | 11
Received Study Intervention | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine + Habit Reversal Training | Placebo + Habit Reversal Training | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 11 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 20
Yale Global Tic Severity Scale Total Tic Score [Mean (Standard Deviation); unit: units on a scale] — The YGTSS is a clinician-administered scale of tic severity. It has two subscale scores of motor tic severity (range: 0-25) and phonic tic severity (range: 0-25) that are summed to produce a total tic score (range: 0-50). Higher total tic scores correspond with greater tic severity.
  units on a scale | 21.89 (6.05) | 18.27 (3.85) | 19.90 (5.16)

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Motor/Vocal Tic Scale (HM/VTS)
Description: Participants can nominate up to five motor and five vocal tics they deem bothersome on the HM/VTS. Each bothersome tic is then rated by a clinician on a 5-point scale ranging from none (0) to severe (4).
  The individual tic scores are summed (minimum of 0 and maximum of 40) and averaged together to create an average tic severity score. Lower scores represent less tic severity, and higher scores indicate greater tic severity.
  The primary outcome will be the difference in the average score of the two bothersome tics on the HM/VTS that were targeted in treatment (range: 0-8). Change scores were calculated by subtracting the average of the two bothersome tics on the HM/VTS at post-treatment from the average of the two bothersome tics on the HM/VTS at the pre-treatment assessment. Positive scores indicate improvement/decrease in targeted tic severity, with negative scores indicating increase in targeted tic severity
Time Frame: Pre-treatment, One Week post-treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | D-cycloserine + Habit Reversal Training | Placebo + Habit Reversal Training
Number analyzed (Participants) | 9 | 10
score on a scale | 1.22 (0.62) | 0.70 (0.54)

ADVERSE EVENTS:
Time Frame: Immediately after therapy session (Visit 2) and 1 week after therapy session (Visit 3)
Description: Adverse events were systematically assessed at Visits 2 and 3 using side effect review form derived from the Safety Monitoring Uniform Report Form (SMURF).
Arm/Group | D-cycloserine + Habit Reversal Training | Placebo + Habit Reversal Training
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 3/9 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine + Habit Reversal Training (N=9) | Placebo + Habit Reversal Training (N=10)
Drowsiness (General disorders) | 1 (1) | 0 (0)
Difficulty Falling Asleep (General disorders) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT02582515/Prot_SAP_000.pdf